CLINICAL TRIAL: NCT06393413
Title: Changchun University of Chinese Medicine
Brief Title: To Explore the Therapeutic Potential of Jiedu Yizhi Formula for Alzheimer 's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changchun University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yunqiang Li, Chief investigator, Changchun University of Chinese Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZDSFYLL2023-0010-01
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Ensure the Legality and Compliance of the Testing Process
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jiedu Yizhi Formula (Experimental): The traditional Chinese medicine treatment group received modified Jiedu Yizhi Formula therapy, with no more than 3 flavors, customized based on syndrome differentiation. The herbal composition included 10g of Coptis chinensis Franch (Huanglian, Ranunculaceae, rhizome), 20g of Alpinia oxyphylla Miq.(Yizhiren, Zingiberaceae, fructus), 10g of Chinemys reevesii(Guibanjiao), 10g of Rheum webbianum (Jiu Dahuang, rhizome), 10g of Cornus officinalis (Shanzhuyu, Cornaceae, fructus), 10g of Pheretima aspergillum (Dilong), and 10g of Oreocome striata (Chuanxiong, Apiaceae, rhizome). 300ml of water decoction juice was prepared from each pair of herbs, and 100ml was taken daily after breakfast and dinner.
  Interventions: Drug: Jiedu Yizhi Formula
- Donepezil Hydrochloride Tablets (Sham Comparator): The Western medicine control group, on the other hand, was administered donepezil hydrochloride (Anlishen 5mg/tablet, from Weicai China Pharmaceutical Co., Ltd.) orally before bedtime at a dosage of 5mg per day. After 4 weeks of treatment, clinical reactions were assessed, and no significant abnormal clinical reactions were observed. Subsequently, the dosage was increased to 10mg per day for maintenance therapy, leading to a total of 24 weeks of continuous treatment. Additionally, both patient groups were provided guidance on actively addressing and managing various risk factors associated with Alzheimer's disease, in conjunction with cognitive behavioral training.
  Interventions: Drug: Donepezil Hydrochloride Tablets

INTERVENTIONS:
Drug: Jiedu Yizhi Formula — Observation after 24 weeks of drug treatment
  Arms: Jiedu Yizhi Formula
Drug: Donepezil Hydrochloride Tablets — Donepezil Hydrochloride Tablets
  Arms: Donepezil Hydrochloride Tablets

SUMMARY:
AD patients who met the inclusion criteria in the encephalopathy clinic and treatment area of the Third Clinical Hospital Affiliated to Changchun University of Traditional Chinese Medicine from December 2022 to December 2023 were collected and randomly divided into traditional Chinese medicine experimental group and western medicine control group. The experimental group was treated with Jiedu Yizhi Formula, and the control group was treated with Donepezil Hydrochloride Tablets ( trade name : Aricept ). The two groups were given AD cognitive behavior training and health education at the same time. The course of treatment was 24 weeks. The Western medicine scale was measured before treatment, 12 weeks after treatment and 24 weeks after treatment to evaluate the effect of drugs on cognitive function and daily living ability.

DETAILED DESCRIPTION:
From December 2022 to December 2023, we conducted a prospective randomized controlled single center study on AD patients exhibiting mild to moderate spleen and kidney deficiency, phlegm turbidity, and obstruction of the orifices. These patients were admitted to the outpatient department and treatment area of the Brain Disease Department at the Third Affiliated Clinical Hospital of Changchun University of Chinese Medicine. Following a comprehensive evaluation, the diagnosis of AD was confirmed. This study was conducted in accordance with the principles of the Helsinki Declaration. The practitioner declares that all procedures follow medical regulations and this study was evaluated and approved by the Ethics Committee of the Third Affiliated Clinical Hospital of Changchun University of Traditional Chinese Medicine. The study was designed based on the observation reports presented in the randomized controlled study of strengthening epidemiology (STROBE).The traditional Chinese medicine treatment group received modified Jiedu Yizhi Formula therapy, with no more than 3 flavors, customized based on syndrome differentiation. The herbal composition included 10g of Coptis chinensis Franch (Huanglian, Ranunculaceae, rhizome), 20g of Alpinia oxyphylla Miq.(Yizhiren, Zingiberaceae, fructus), 10g of Chinemys reevesii(Guibanjiao), 10g of Rheum webbianum (Jiu Dahuang, rhizome), 10g of Cornus officinalis (Shanzhuyu, Cornaceae, fructus), 10g of Pheretima aspergillum (Dilong), and 10g of Oreocome striata (Chuanxiong, Apiaceae, rhizome). 300ml of water decoction juice was prepared from each pair of herbs, and 100ml was taken daily after breakfast and dinner. The Western medicine control group, on the other hand, was administered donepezil hydrochloride (Anlishen 5mg/tablet, from Weicai China Pharmaceutical Co., Ltd.) orally before bedtime at a dosage of 5mg per day. Subsequently, the dosage was increased to 10mg per day for maintenance therapy, leading to a total of 24 weeks of continuous treatment. Additionally, both patient groups were provided guidance on actively addressing and managing various risk factors associated with Alzheimer's disease, in conjunction with cognitive behavioral training.

ELIGIBILITY:
Inclusion Criteria:

(1) Meet the above NIA-AA AD diagnostic criteria; (2) Meets the diagnostic criteria for traditional Chinese medicine syndromes mentioned above; (3) Age range from 55 to 85 years old, regardless of gender; (4) MMSE scale scores range from 10 to 26 points; (5) The CDR scale scores 1 or 2 points; (6) The HAMD scale score is less than 8 points; (7) HAMA scale score below 7 points; (8) At least 4 elements of kidney deficiency, spleen deficiency, marrow deficiency, blood stasis, and phlegm turbidity syndrome in the PES-D/11 scale score are valid, and may be accompanied by toxic excess syndrome elements (the sum of scores greater than or equal to 7 points is considered valid); (9) HIS scale score below 5 points; (10) Family members agree and sign an informed consent form.

Exclusion Criteria:

(1) Severe dementia patients; (2) Other types of dementia such as vascular dementia, frontotemporal lobe dementia, Lewy body dementia, mixed dementia, as well as secondary dementia caused by infection, poisoning, metabolism, tumors, and other reasons; (3) There are other diseases that may cause cognitive impairment; (4) Patients who cannot fully cooperate with the assessment; (5) Patients with unstable vital signs and critical condition; (6) Patients with concomitant psychiatric disorders; (7) Patients with scores of less than 7 on the PES-D/11 scale for spleen deficiency, kidney deficiency, marrow deficiency, blood stasis, and phlegm turbidity; (8) Patients with long-term alcohol or drug abuse that affects efficacy evaluation; (9) Patients who have experienced serious adverse reactions or allergies to the drugs in this study due to previous use of traditional Chinese medicine.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Mini-mental State Examination(MMSE) | 24 weeks
  The most widely used cognitive screening tool in the world today, the MMSE was created by Folstein et al. in 1975. It is frequently used to measure endpoint outcomes, evaluate cognitive levels, and screen for cognitive impairment. 30 points is the highest score, and 0 points is the lowest. The better the cognitive function, the higher the score.
Montreal Cognitive Assessment (MoCA) | 24 weeks
  Professor Nasreddine and colleagues created MoCA in 2004. Recall, naming, abstraction, language, attention, visual spatial and executive abilities, and directional abilities are among the eight areas on the scale that assess cognitive performance. Higher scores indicate stronger cognitive function. The scores range from 0 to 30.
Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-cog） | 24 weeks
  The 12-item ADAS cog is used to evaluate the degree of memory, language, and other cognitive impairments in people with Alzheimer's disease. Of them, four evaluate language, five evaluate memory and direction, two evaluate practical competence, and one evaluate focus and attention. The more severe the cognitive impairment, the higher the score on the ADAS log, which ranges from 0 to 70 points. The better the therapeutic impact, the lower the score after taking medication.
Clinical dementia rating(CDR) | 24 weeks
  CDR (Clinical Dementia Rating) is a standard for evaluating the degree of dementia, which includes a series of cognitive function assessments, including memory, attention, understanding, sense of direction, computational ability, etc. The evaluation results include 0 points, 0.5 points, 1 point, 2 points, 3 points, 0 points indicating normal, and 0.5 points indicating mild dementia,
  1 point represents moderate dementia, 2 points represents severe dementia, and 3 points represents terminal dementia.

SECONDARY OUTCOMES:
Activity of daily living（ ADL ） | 24 weeks
  Activity of daily life refers to the necessary activities that a person engages in every day to meet their daily needs, including eating, dressing, washing, bathing, toileting, dressing, etc. Functional movements include turning over, sitting up from bed, transferring, walking, driving a wheelchair, going up and down stairs, etc. The score ranges from 0 to 100 points, and the higher the score, the stronger the daily living ability.
Hamilton Depression Stable （HAMD ） | 24 weeks
  Evaluate mental state using the HAMD scale.During the diagnosis and treatment process, it was found that many AD patients are accompanied by varying degrees of depression, which will also affect the improvement of their cognitive function. In terms of efficacy evaluation indicators, in addition to evaluating cognitive function scales, HAMD should also be included in the observation indicators. The score range for each scoring item is 0-4 points, with a total score of 0-76 points. When scoring, the doctor or evaluator needs to select the scoring item that best matches the symptoms of the evaluated person based on their actual situation, and give corresponding scores. The higher the score, the more severe the depressive symptoms are.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Dr., Study Director — Affiliated Hospital
Locations (1):
- Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR